CLINICAL TRIAL: NCT02628899
Title: Feasibility of Transcatheter Aortic Valve Replacement in Low-Risk Patients With Symptomatic, Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Low Risk TAVR
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Prospective TAVR Arm (Other): 200 patients prospectively undergoing transfemoral TAVR
  Interventions: Device: Transfemoral TAVR
- Historical SAVR Controls (Other): Historical controls will be selected from among patients at the same site who have undergone isolated bioprosthetic SAVR within the previous 36 months. TAVR patients will then be matched to SAVR patients using STS database variables to perform propensity matching, including (but not limited to) age, gender, race, ethnicity, STS score, and valve prosthesis size.
  Interventions: Device: SAVR
- Low-Risk TAVR with Bicuspid Aortic Valve (Other): The third arm of the trial will comprise a registry of TAVR in up to 100 low-risk patients with bicuspid aortic valve. The results from the registry arm will be analyzed independently.
  Interventions: Device: Transfemoral TAVR

INTERVENTIONS:
Device: Transfemoral TAVR
  Other Names: Transcatheter aortic valve replacement
  Arms: Low-Risk TAVR with Bicuspid Aortic Valve; Prospective TAVR Arm
Device: SAVR
  Other Names: Surgical Aortic Valve Replacement
  Arms: Historical SAVR Controls

SUMMARY:
To assess the safety and feasibility of Transcatheter Aortic Valve Replacement (TAVR) with commercially available bioprostheses in patients with severe, symptomatic aortic stenosis (AS) who are low-risk (STS score ≤3%) for surgical aortic valve replacement (SAVR).

DETAILED DESCRIPTION:
Trial Objectives: To assess the safety and feasibility of Transcatheter Aortic Valve Replacement (TAVR) with commercially available bioprostheses in patients with severe, symptomatic aortic stenosis (AS) who are low-risk (STS score ≤3%) for surgical aortic valve replacement (SAVR).

Methodology: This is a multicenter, prospective trial of TAVR in low-risk patients at up to twelve sites in the United States. The trial will have three arms. The first will comprise 200 patients undergoing transfemoral TAVR. The second arm will comprise200 closely matched historical controls who underwent isolated bioprosthetic SAVR.

Historical controls will be selected from among patients at the same site who have undergone isolated bioprosthetic SAVR within the previous 36 months. TAVR patients will then be matched to SAVR patients using STS database variables to perform propensity matching, including (but not limited to) age, gender, race, ethnicity, STS score, and valve prosthesis size. Once the historical matched controls are identified, detailed chart review will abstract in-hospital and 30-day outcomes for the SAVR cohort.

The third arm of the trial will comprise a registry of TAVR in up to 100 low-risk patients with bicuspid aortic valve. The results from the registry arm will be analyzed independently.

Primary Efficacy Endpoint: All-cause mortality at 30 days following transfemoral TAVR vs. bioprosthetic SAVR.

Primary Safety Endpoint: Defined as the composite of major adverse events at 30 days:

a. all-cause mortality c. spontaneous myocardial infarction (MI) d. reintervention: defined as any cardiac surgery or percutaneous reintervention that repairs, alters, or replaces a previously implanted aortic valve e. VARC life-threatening bleeding f. Increase in serum creatinine to ≥300% (>3x increase compared to baseline) OR serum creatinine ≥4.0 mg/dL with an acute increase ≥0.5 mg/dL OR new requirement for dialysis g. coronary artery obstruction requiring percutaneous or surgical intervention h. VARC major vascular complication i. cardiac tamponade j. cardiac perforation k. pericarditis l. mediastinitis m. hemolysis n. infective endocarditis o. moderate or severe aortic insufficiency p. significant aortic stenosis q. permanent pacemaker implantation r. new-onset atrial fibrillation

Secondary Endpoints (TAVR Cohort):

1. Major adverse cardiovascular and cerebrovascular events (MACCE) at 30 days, 6 months, 12 months, and 2, 3, 4 and 5 years, defined as the composite of:

   1. all-cause mortality
   2. stroke
   3. spontaneous MI
   4. reintervention
2. The occurrence of the individual components of MACCE at 30 days, 6 months, 12 months, and 2, 3, 4, and 5 years (including stoke).
3. The composite of major adverse device events post-procedure, and at 6 months, 1 year, and 2, 3, 4, 5 years
4. VARC major vascular complications, at 30 days and 1 year
5. VARC life-threatening or disabling bleeding, at 30 days and 1 year
6. Technical success upon exit from the operating room or catheterization laboratory, defined as all of the following:

   1. alive
   2. successful access, delivery, and retrieval of the device and/or delivery system
   3. correct positioning and successful deployment of the valve
   4. no need for unplanned or emergency surgery or reintervention related to the device or access procedure, including reinstitution of cardiopulmonary bypass post-weaning for SAVR patients
7. Device success at 30 days and 1 year, defined as all of the following:

   1. absence of procedural mortality
   2. correct positioning of a single prosthetic heart valve in the proper anatomical location
   3. device performing as intended:

1. No migration, erosion, embolization, detachment, fracture, hemolysis requiring transfusion, thrombosis, or endocarditis 2. Intended performance of the heart valve: no prosthesis-patient mismatch, mean aortic valve gradient <20 mm Hg OR peak velocity <3 m/s, AND no moderate or severe bioprosthetic valve regurgitation 8. Procedural success at 30 days, defined as device success AND no major adverse device events 9. Bioprosthetic valve regurgitation, defined as either moderate or severe aortic regurgitation OR moderate or severe paravalvular leak, at hospital discharge, 12 months, and 2, 3, 4, and 5 years 10. Incidence of new-onset atrial fibrillation at hospital discharge, and at 30 days, 12 months, and 2, 3, 4, and 5 years.

11. Conduction disturbance requiring permanent pacemaker implantation at hospital discharge, 12 months, and 2, 3, 4, and 5 years.

12. Change in NYHA class from baseline to 30 days, baseline to 6 months, baseline to 12 months, and baseline to 2-5 years.

13. Change in distance walked during 6-minute walk test from baseline to 12 months.

14. Change in responses to the short form Kansas City Cardiomyopathy Questionnaire (KCCQ-12) from baseline to 12 months.

15. Echocardiographic assessment of the bioprosthetic valve post-procedure, at 12 months, and at years 2-5, including (but not limited to):

a. aortic valve mean gradient, maximum gradient, and peak velocity b. calculated aortic valve area c. degree of bioprosthetic valve regurgitation 16. Assessment for subclinical leaflet thrombosis with multislice computed tomography, or transesophageal echocardiography if GFR <50 mL/min/m2, at 1 to 2 months.

17. Individual patient level Success all of the following and device success:

1. No re-hospitalizations or re-interventions for the underlying condition (e.g., HF)
2. Return to prior living arrangement (or equivalent)
3. Improvement vs. baseline in symptoms (NYHA Class decrease ≥ 1)
4. Improvement vs. baseline in functional status (6MWT increase ≥ 50 meters)
5. Improvement vs. baseline in QoL (KCCQ increase ≥ 10)

Number of Trial Sites: 12

Sample Size: 200 consecutive patients and 200 historical controls, and an additional 100 (up to) patients with bicuspid aortic valve

Patient Population: Patients with severe, symptomatic AS who are determined by the Heart Team to be at low surgical risk (STS score ≤3%).

ELIGIBILITY:
Inclusion Criteria:

1. Severe, degenerative AS, defined as:

   1. mean aortic valve gradient ≥40 mm Hg OR Vmax ≥4 m/sec AND
   2. calculated aortic valve area ≤1.0 cm2 OR aortic valve area index ≤0.6 cm2/m2
2. Symptomatic AS, defined as a history of at least one of the following:

   1. dyspnea that qualifies at New York Heart Association (NYHA) class II or greater
   2. angina pectoris
   3. cardiac syncope
3. The Heart Team, including at least one cardiothoracic surgeon and one interventional cardiologist, deem the patient to be reasonable for transfemoral TAVR with a commercially available bioprosthetic valve
4. The Heart Team agrees that the patient is low-risk, quantified by an estimated risk of ≤3% by the calculated STS score for operative mortality at 30 days; AND agrees that SAVR would be an appropriate therapy if offered.
5. The Heart Team agrees that transfemoral TAVR is anatomically feasible, based upon multislice CT measurements
6. Procedure status is elective
7. Expected survival is at least 24 months

   For the bicuspid cohort only:
8. Aortic Stenosis of a bicuspid aortic valve

Exclusion Criteria:

1. Concomitant disease of another heart valve or the aorta that requires either transcatheter or surgical intervention
2. Any condition that is considered a contraindication for placement of a bioprosthetic aortic valve (e.g. patient requires a mechanical aortic valve)
3. Aortic stenosis secondary to a bicuspid aortic valve (except for the bicuspid valve cohort)
4. Prior bioprosthetic surgical aortic valve replacement
5. Mechanical heart valve in another position
6. End-stage renal disease requiring hemodialysis or peritoneal dialysis, or a creatinine clearance <20 cc/min
7. Left ventricular ejection fraction <20%
8. Recent (<6 months) history of stroke or transient ischemic attack
9. Symptomatic carotid or vertebral artery disease, or recent (<6 weeks) surgical or endovascular treatment of carotid stenosis
10. Any contraindication to oral antiplatelet or anticoagulation therapy following the procedure, including recent or ongoing bleeding, or HASBLED score >3
11. Severe coronary artery disease that is unrevascularized
12. Recent (<30 days) acute myocardial infarction
13. Patient cannot undergo transfemoral TAVR for anatomic reasons (as determined by supplemental imaging studies); this would include inadequate size of iliofemoral access vessels or an aortic annulus size that is not accommodated by the commercially available valves
14. Any comorbidity not captured by the STS score that would make SAVR high risk, as determined by a cardiothoracic surgeon who is a member of the heart team; this includes:

    1. porcelain or severely atherosclerotic aorta
    2. frailty
    3. hostile chest
    4. IMA or other conduit either crosses midline of sternum or is adherent to sternum
    5. severe pulmonary hypertension (PA systolic pressure > 2/3 of systemic pressure)
    6. severe right ventricular dysfunction
15. Ongoing sepsis or infective endocarditis
16. Recent (<30 days) or ongoing bleeding that would preclude treatment with anticoagulant or antiplatelet therapy, including recent gastrointestinal bleeding
17. Uncontrolled atrial fibrillation (resting heart rate >120 beats per minute)
18. Severe chronic obstructive pulmonary disease, as demonstrated by forced expiratory volume (FEV1) <750 cc
19. Liver failure with Childs class C or D
20. Pre-procedure shock, inotropes, mechanical assist device, or cardiac arrest
21. Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures
22. Known allergy to warfarin or aspirin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at 30 days following transfemoral TACR vs. bioprosthetic SAVR | 30 days following transfemoral TAVR vs. bioprosthetic SAVR
  All-cause mortality at 30 days following transfemoral TACR vs. bioprosthetic SAVR
Composite of major adverse events at 30 days | 30 days
  Composite of major adverse events at 30 days
  1. all-cause mortality
  2. stroke
  3. spontaneous myocardial infarction (MI)
  4. reintervention: defined as any cardiac surgery or percutaneous reintervention that repairs, alters, or replaces a previously implanted aortic valve
  5. VARC life-threatening bleeding
  6. Increase in serum creatinine to ≥300% (>3x increase compared to baseline) OR serum creatinine ≥4.0 mg/dL with an acute increase ≥0.5 mg/dL OR new requirement for dialysis
  7. coronary artery obstruction requiring percutaneous or surgical intervention
  8. VARC major vascular complication
  9. cardiac tamponade
  10. cardiac perforation
  11. pericarditis
  12. mediastinitis
  13. hemolysis
  14. infective endocarditis
  15. moderate or severe aortic insufficiency
  16. significant aortic stenosis
  17. permanent pacemaker implantation
All Cause Mortality | 30 days
All Stroke (disabling and non-disabling, ischemic and hemorrhagic | 30 Days
Life Threatening and Major Bleeding | 30 days
Major Vascular Complications | 30 days
Hospitalizations for valve-related symptoms or worsening congestive heart failure | 30 days

SECONDARY OUTCOMES:
composite of all-cause mortality, stroke, spontaneous MI, re-intervention | 30 days, 6 months, 12 months, and 2,3,4 and 5 years
  composite of:
  1. all-cause mortality
  2. stroke
  3. spontaneous MI
  4. re-intervention 2. The occurrence of the individual components of MACCE at 30 days, 6 months, 12 months, and 2, 3, 4, and 5 years. 3. The composite of major adverse device events post-procedure, and at 6 months, 1 year, and 2, 3, 4, 5 years 4. VARC major vascular complications, at 30 days and 1 year 5. VARC life-threatening or disabling bleeding, at 30 days and 1 year 6. Assessment for subclinical leaflet thrombosis with multislice computed tomography, or transesophageal echocardiography if GFR <50 mL/min/m2, at 1 to 2 months.
VARC - 2 Device Success | 30 days
  Absence of procedural mortality AND Correct positioning of a single prosthetic heart valve into the proper anatomical location AND Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient<20 mm Hg or peak velocity<3 m/s, AND no moderate or severe prosthetic valve regurgitation)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Sutter Health System, Sacramento, California
  - Foundation for Cardiovascular Medicine, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Maine Medical Center, Portland, Maine
  - The Valley Hospital, Ridgewood, New Jersey
  - Stony Brook Hospital, Stony Brook, New York
  - St. John Health System, Tulsa, Oklahoma
  - Miriam Hospital, Providence, Rhode Island
  - Henrico Doctors' Hospital, Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia

REFERENCES:
- [Background] Waksman R, Rogers T, Torguson R, Gordon P, Ehsan A, Wilson SR, Goncalves J, Levitt R, Hahn C, Parikh P, Bilfinger T, Butzel D, Buchanan S, Hanna N, Garrett R, Asch F, Weissman G, Ben-Dor I, Shults C, Bastian R, Craig PE, Garcia-Garcia HM, Kolm P, Zou Q, Satler LF, Corso PJ. Transcatheter Aortic Valve Replacement in Low-Risk Patients With Symptomatic Severe Aortic Stenosis. J Am Coll Cardiol. 2018 Oct 30;72(18):2095-2105. doi: 10.1016/j.jacc.2018.08.1033. Epub 2018 Aug 28. PMID 30170075
- [Background] Waksman R, Corso PJ, Torguson R, Gordon P, Ehsan A, Wilson SR, Goncalves J, Levitt R, Hahn C, Parikh P, Bilfinger T, Butzel D, Buchanan S, Hanna N, Garrett R, Buchbinder M, Asch F, Weissman G, Ben-Dor I, Shults C, Bastian R, Craig PE, Ali S, Garcia-Garcia HM, Kolm P, Zou Q, Satler LF, Rogers T. TAVR in Low-Risk Patients: 1-Year Results From the LRT Trial. JACC Cardiovasc Interv. 2019 May 27;12(10):901-907. doi: 10.1016/j.jcin.2019.03.002. Epub 2019 Mar 12. PMID 30860059
- [Background] Khan JM, Rogers T, Waksman R, Torguson R, Weissman G, Medvedofsky D, Craig PE, Zhang C, Gordon P, Ehsan A, Wilson SR, Goncalves J, Levitt R, Hahn C, Parikh P, Bilfinger T, Butzel D, Buchanan S, Hanna N, Garrett R, Shults C, Garcia-Garcia HM, Kolm P, Satler LF, Buchbinder M, Ben-Dor I, Asch FM. Hemodynamics and Subclinical Leaflet Thrombosis in Low-Risk Patients Undergoing Transcatheter Aortic Valve Replacement. Circ Cardiovasc Imaging. 2019 Dec;12(12):e009608. doi: 10.1161/CIRCIMAGING.119.009608. Epub 2019 Dec 12. PMID 31826675
- [Background] Rogers T, Torguson R, Bastian R, Corso P, Waksman R. Feasibility of transcatheter aortic valve replacement in low-risk patients with symptomatic severe aortic stenosis: Rationale and design of the Low Risk TAVR (LRT) study. Am Heart J. 2017 Jul;189:103-109. doi: 10.1016/j.ahj.2017.03.008. Epub 2017 Mar 14. PMID 28625366
- [Derived] Reddy P, Rodriguez-Weisson FJ, Medranda GA, Merdler I, Cellamare M, Gordon P, Ehsan A, Parikh P, Bilfinger T, Buchbinder M, Roberts D, Hanna N, Ben-Dor I, Satler LF, Garcia-Garcia HM, Asch FM, Weissman G, Sadeghpour A, Schults CC, Waksman R, Rogers T. Impact of Calcified Raphe on TAVR in Bicuspid Patients: Predicting Redo-TAVR Feasibility and Virtual Planning Implications. Circ Cardiovasc Interv. 2025 Jun;18(6):e014802. doi: 10.1161/CIRCINTERVENTIONS.124.014802. Epub 2025 Apr 22. PMID 40260550
- [Derived] Bhogal S, Waksman R, Shea C, Zhang C, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Weissman G, Ben-Dor I, Shults CC, Ali S, Garcia-Garcia HM, Satler LF, Rogers T. Self-expanding and balloon-expandable valves in low risk TAVR patients. Int J Cardiol. 2024 Jan 15;395:131431. doi: 10.1016/j.ijcard.2023.131431. Epub 2023 Oct 12. PMID 37832606
- [Derived] Waksman R, Bhogal S, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Kim FY, Weissman G, Ben-Dor I, Shults CC, Ali S, Sutton JA, Shea C, Zhang C, Garcia-Garcia HM, Satler LF, Rogers T. Transcatheter Aortic Valve Replacement and Impact of Subclinical Leaflet Thrombosis in Low-Risk Patients: LRT Trial 4-Year Outcomes. Circ Cardiovasc Interv. 2023 May;16(5):e012655. doi: 10.1161/CIRCINTERVENTIONS.122.012655. Epub 2023 May 16. PMID 37192308
- [Derived] Medranda GA, Soria Jimenez CE, Torguson R, Case BC, Forrestal BJ, Ali SW, Shea C, Zhang C, Wang JC, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Weissman G, Shults CC, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R, Rogers T. Lifetime management of patients with symptomatic severe aortic stenosis: a computed tomography simulation study. EuroIntervention. 2022 Aug 5;18(5):e407-e416. doi: 10.4244/EIJ-D-21-01091. PMID 35321859
- [Derived] Medranda GA, Rogers T, Forrestal BJ, Case BC, Yerasi C, Chezar-Azerrad C, Shults CC, Torguson R, Shea C, Parikh P, Bilfinger T, Cocke T, Brizzio ME, Levitt R, Hahn C, Hanna N, Comas G, Mahoney P, Newton J, Buchbinder M, Zhang C, Craig PE, Weigold WG, Asch FM, Weissman G, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R. Balloon-Expandable Valve Geometry After Transcatheter Aortic Valve Replacement in Low-Risk Patients With Bicuspid Versus Tricuspid Aortic Stenosis. Cardiovasc Revasc Med. 2021 Dec;33:7-12. doi: 10.1016/j.carrev.2021.03.027. Epub 2021 Apr 6. PMID 34078581
- [Derived] Waksman R, Torguson R, Medranda GA, Shea C, Zhang C, Gordon P, Ehsan A, Wilson SR, Levitt R, Hahn C, Parikh P, Bilfinger T, Butzel D, Buchanan S, Hanna N, Buchbinder M, Asch F, Weissman G, Ben-Dor I, Shults C, Garcia-Garcia HM, Satler LF, Rogers T. Transcatheter aortic valve replacement in low-risk patients: 2-year results from the LRT trial. Am Heart J. 2021 Jul;237:25-33. doi: 10.1016/j.ahj.2021.03.006. Epub 2021 Mar 10. PMID 33713618
- [Derived] Khan JM, Rogers T, Weissman G, Torguson R, Rodriguez-Weisson FJ, Chezar-Azerrad C, Greenspun B, Gupta N, Medvedofsky D, Zhang C, Gordon P, Ehsan A, Wilson SR, Goncalves J, Levitt R, Hahn C, Parikh P, Bilfinger T, Butzel D, Buchanan S, Hanna N, Garrett R, Shults C, Buchbinder M, Garcia-Garcia HM, Kolm P, Satler LF, Hashim H, Ben-Dor I, Asch FM, Waksman R. Anatomical Characteristics Associated With Hypoattenuated Leaflet Thickening in Low-Risk Patients Undergoing Transcatheter Aortic Valve Replacement. Cardiovasc Revasc Med. 2021 Jun;27:1-6. doi: 10.1016/j.carrev.2020.09.034. Epub 2020 Sep 25. PMID 33129688
- [Derived] Waksman R, Craig PE, Torguson R, Asch FM, Weissman G, Ruiz D, Gordon P, Ehsan A, Parikh P, Bilfinger T, Levitt R, Hahn C, Roberts D, Ingram M, Hanna N, Comas G, Zhang C, Ben-Dor I, Satler LF, Garcia-Garcia HM, Shults C, Rogers T. Transcatheter Aortic Valve Replacement in Low-Risk Patients With Symptomatic Severe Bicuspid Aortic Valve Stenosis. JACC Cardiovasc Interv. 2020 May 11;13(9):1019-1027. doi: 10.1016/j.jcin.2020.02.008. Epub 2020 Feb 24. PMID 32381181
- [Derived] Ozaki Y, Garcia-Garcia HM, Rogers T, Torguson R, Craig PE, Hideo-Kajita A, Gordon P, Ehsan A, Parikh P, Bilfinger T, Butzel D, Buchanan S, Levitt R, Hahn C, Buchbinder M, Hanna N, Garrett R, Wilson SR, Goncalves JA, Ali S, Asch FM, Weissman G, Shults C, Ben-Dor I, Satler LF, Waksman R. Coronary Artery Disease Assessed by Computed Tomography-Based Leaman Score in Patients With Low-Risk Transcatheter Aortic Valve Implantation. Am J Cardiol. 2020 Apr 15;125(8):1216-1221. doi: 10.1016/j.amjcard.2020.01.022. Epub 2020 Jan 28. PMID 32087995